CLINICAL TRIAL: NCT04700917
Title: Internet-Based Cognitive Behavioural Program for Managing Stress With Inflammatory Bowel Disease: A Randomized Controlled Trial
Brief Title: Internet-Based Cognitive Behavioural Program for Managing Stress With IBD: An RCT
Acronym: iCBT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Patricia Furer, Associate Professor, University of Manitoba
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H2020:430
Record Dates: First submitted 2021-01-06; First posted 2021-01-08 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Inflammatory Bowel Diseases; Anxiety; Depression; Stress
Keywords: Inflammatory Bowel Disease, Anxiety, Depression, Stress, Online Intervention
MeSH Terms: conditions — Inflammatory Bowel Diseases; Anxiety Disorders; Depression | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): This group will receive the iCBT for IBD online intervention once enrolled.
  Interventions: Behavioral: Cognitive Behavioural Therapy
- Treatment as Usual (No Intervention): This group will be offered the iCBT for IBD intervention 24 weeks after enrollment.

INTERVENTIONS:
Behavioral: Cognitive Behavioural Therapy — Internet-Based CBT
  Arms: Intervention Group

SUMMARY:
The study will examine the efficacy of an internet-based cognitive behavioural therapy (iCBT) for Inflammatory Bowel Disease (IBD) intervention to reduce stress, anxiety, and depression in individuals with IBD and comorbid clinically elevated t anxiety and/or depressive symptoms. The investigators will conduct a two-arm RCT comparing participants receiving the iCBT intervention (intervention group) and those receiving Treatment As Usual (TAU).

DETAILED DESCRIPTION:
Inflammatory bowel disease (IBD) affects over a quarter of a million Canadians and this rate is expected to increase to 403,000 by year 2030 (Kaplan, Bernstein, Coward, Bitton, Murthy, Nguyen, Lee, Cooke-Lauder, Benchimol, 2019). The disease has a high burden for patients, with unpredictable, painful symptoms often requiring costly medications and surgery to facilitate disease remission. It is well established that individuals with IBD have significantly higher rates of anxiety and depression compared to the general population. (Bernstein, 2017; Graff, Walker, & Bernstein, 2009; Mikocka-Walus, Knowles, Keefer, Graff, 2016; Walker, Ediger, Graff, Greenfeld, Clara, Lix, Rawsthorne, Miller, Rogala, McPhail, & Bernstein, 2008).

There is growing research on psychological treatment for individuals with IBD, providing some evidence that Cognitive Behavioural Therapy (CBT) reduces psychological distress in this population (Knowles, Monshat, & Castle, 2013). Traditional CBT delivery methods involve in-person treatment, with multiple sessions over time, either one-on-one or in small groups. Development of alternate modes of effective treatment delivery is vital to enhance access and facilitate availability, particularly given limited mental health service availability. Internet-Based Cognitive Behaviour Therapy (iCBT) may be an effective alternative treatment for persons with IBD and related stress, anxiety and/or depression (McCombie, 2016) as it may mitigate the aforementioned challenges. Potential benefits of iCBT include enhanced cost effectiveness, little to no wait time to begin treatment, and increased accessibility.

Our research group developed and pilot-tested an internet-based cognitive behavioural therapy (iCBT) intervention targeting stress, anxiety and/or depression in adults with IBD. The intervention is housed on the Minddistrict online platform, the same platform used in our pilot study (HREB Ethics HS22087 (H2018:333) (Minddistrict, 2018, June, 1).The program was designed to be completed over 12 weeks. The study coordinator will be tracking participants' progress through the intervention by reviewing completion of questionnaires and modules.

The intervention includes 9 core modules and 3 optional modules. CORE Modules: 1. About the program, 2. IBD and Stress, 3. Relaxation Strategies, 4, Commitment to Living Life Fully, 5. The Brain-Gut Connection, 6. Understanding Anxiety, 7. Overcoming Avoidance, 8. Depression, 9. Behavioural Activation Optional Modules: 11. IBD and the Workplace, 12. Coping with Pain through Mindfulness, 13. Fatigue and Sleep

The next stage in extending this research is to conduct a randomized control trial (RCT) to determine the efficacy of this internet-based intervention, utilizing a control condition and ensuring adequate sample size powered to detect differences between the intervention group and Treatment as Usual (TAU).

Participants will be adults with confirmed inflammatory bowel disease, recruited from local enrollees of the IMAGINE study described earlier (IMAGINE, 2020, July, 2). They will be contacted by email to invite for participation in this study.

Participants will be randomized using a computer-generated randomization schedule which allows for allocation concealment with a ratio of 1.2 (iCBT) : 1.0 (TAU).

ELIGIBILITY:
Inclusion Criteria:

* Participants will need to be at least 18 years of age or older, be diagnosed by a physician with IBD (Crohn's disease or Ulcerative Colitis), have anxiety and/or depression scores > 8 on the Hospital Anxiety and Depression Scale (HADS-A or HADS-D), have access to a computer, and be literate in the English language. Participants may be on psychotropic medication but dosage should be stable for at least six weeks prior to study enrollment.

Exclusion Criteria:

* Individuals who have had, within the last six months, suicidal ideation or suicidal intent, self-harming behaviour, active substance use disorder, psychotic disorder, or an eating disorder will be excluded. Presence of these behaviours and disorders will be determined through the screening process described in the next section. Individuals who are currently receiving cognitive behavioral treatment for an anxiety or mood disorder, or have participated in such treatment in the previous three months, are not eligible for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 352 (Estimated)
Dates: Start 2021-03-16 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
PSS-4 | Baseline, 6, 12 and 24 weeks
  Change in Perceived Stress Scale 4 (PSS-4) scale measuring psychological stress (4 items); likert scale 0 (never) to 4 (very often); higher scores indicate higher levels of perceived stress
HADS | Baseline, 6, 12 and 24 weeks
  Change in Hospital Anxiety and Depression Scale (HADS) scale measuring anxiety and depression (14 items); likert scale 0 (not at all) to 3 (most of the time); higher scores(summed) indicate presence of anxiety or depression

SECONDARY OUTCOMES:
PROMIS-29 | Baseline, 6, 12 and 24 weeks
  Change in Patient-Reported Outcomes Measurement Information System - 29 (PROMIS-29) scale measuring health-related quality of life (29 items); likert scale 1 to 5, varying anchor points; in symptom oriented domains higher scores represent worse symptomology and in function oriented domains higher scores represent better functioning
WSAS | Baseline, 6, 12 and 24 weeks
  Change in the Work and Social Adjustment Scale (WSAS) scale measuring how inflammatory bowel disease impact daily functioning; likert scale 1(not at all) to 5 (very severely); higher scores indicate higher levels higher functional impairment
IBDSI-SF | Baseline, 6, 12 and 24 weeks
  Change in Inflammatory Bowel Disease Symptom Inventory - Short Form (IBDSI) scale measuring symptoms of inflammatory bowel disease; likert scale with varying anchor points
CGI | Baseline, 6,12 and 24 weeks
  Change in Clinical Global Impression - Improvement scale (CGI-I) scale measuring confidence in ability to manage stress (2 items); likert scale with varying anchor points; higher scores indicate higher stress and lower confidence

CONTACTS AND LOCATIONS:
Locations (1):
- University of Manitoba, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tiles-Sar N, Neuser J, de Sordi D, Baltes A, Preiss JC, Moser G, Timmer A. Psychological interventions for treatment of inflammatory bowel disease. Cochrane Database Syst Rev. 2025 Apr 17;4(4):CD006913. doi: 10.1002/14651858.CD006913.pub3. PMID 40243391